CLINICAL TRIAL: NCT04235114
Title: Evaluation of 89Zr-DFO-nimotuzumab for Non-invasive Imaging of EGFR Positive Cancers by Positron Emission Tomography (PET)
Brief Title: Evaluation of 89Zr-DFO-nimotuzumab for Non-invasive Imaging of EGFR+ Cancers by Positron Emission Tomography (PET)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Rajan Rakheja, Clinical Assistant Professor, University of Saskatchewan
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: Bio 17-288
Record Dates: First submitted 2018-10-13; First posted 2020-01-21 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer; Colorectal Cancer
Keywords: 89Zr; Nimotuzumab; Lung cancer; Colorectal cancer; EGFR; PET; PET/CT; Imaging; 89Zr-DFO-nimotuzumab
MeSH Terms: conditions — Lung Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single center, open-label, phase I/II diagnostic imaging study to assess the diagnostic quality of 89Zr-DFO-nimotuzumab with PET.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Establish Imaging Time (Experimental): Participants will receive an i.v. injection of 50 mg 2 mCi 89Zr-DFO-nimotuzumab. Participants will undergo imaging at four different time points till day 7 after infusion. Vitals, blood sample and urine sample will be collected every time before imaging. Participants will be followed up for any adverse event until day 30 post administration
  Interventions: Drug: 50 mg 89Zr-DFO-Nimotuzumab
- Diagnostic Quality (Experimental): Participants will receive an i.v. injection of 50 mg 2 mCi 89Zr-DFO-nimotuzumab. Participants will undergo imaging once at the best time calculated from arm 1 participants. Vitals, blood sample and urine sample will be collected before imaging. Participants will be followed up for any adverse event until day 30 post administration
  Interventions: Drug: 50 mg 89Zr-DFO-Nimotuzumab
- Establish Cold Dose (Experimental): Participants will receive an i.v. injection of 1 mg 2 mCi 89Zr-DFO-nimotuzumab. Participants will undergo imaging at four different time points till day 7 after infusion. Vitals, blood sample and urine sample will be collected every time before imaging. Participants will be followed up for any adverse event until day 30 post administration
  Interventions: Drug: 1 mg 89Zr-DFO-Nimotuzumab

INTERVENTIONS:
Drug: 50 mg 89Zr-DFO-Nimotuzumab — A maximum of 2 mCi (range 1 - 2 mCi) 50 mg of 89Zr-DFO-nimotuzumab will be injected intravenously over a period of at 2 - 3 minutes. Injection will be followed by a normal saline flush of 20-30 mL. PET/CT scan will be done at different time points post infusion.
  Arms: Diagnostic Quality; Establish Imaging Time
Drug: 1 mg 89Zr-DFO-Nimotuzumab — A maximum of 2 mCi (range 1 - 2 mCi) 1 mg of 89Zr-DFO-nimotuzumab will be injected intravenously over a period of at 2 - 3 minutes. Injection will be followed by a normal saline flush of 20-30 mL. PET/CT scan will be done at different time points post infusion.
  Arms: Establish Cold Dose

SUMMARY:
Over-expression of Epidermal Growth Factor Receptor (EGFR) on cells occurs in all aggressive cancers of epithelial origin. Existing tests for monitoring EGFR expression are invasive and not reliable. There needs to be a better way to measure EGFR expression in cancerous tumors to better tailor cancer treatments.

This clinical trial aims to demonstrate the feasibility of imaging cancers that express EGFR using 89Zr-DFO-nimotuzumab and Positron Emission Tomography (PET)/Computerized Tomography (CT). By non-invasively imaging the status of EGFR, 89Zr-DFO-nimotuzumab could be used to assist in the identification of patients who are likely to respond to anti-EGFR treatments, including nimotuzumab. The hypothesis is that 89Zr-DFO-nimotuzumab will accumulate to tumors over-expressing EGFR making them visible when imaged with PET/CT. This hypothesis will be tested in this study, along with the optimal imaging time and diagnostic ability.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 80 years old.
* EGFR-positive cancer defined by a board certified pathologist
* Primary or metastatic lesion size >= 1.5 cm as determined by imaging studies (ultrasonography, mammography, CT or MRI) or physical examination.
* Able to give informed consent.
* Not currently pregnant or nursing: If female subject must be surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), post-menopausal (cessation of menses for > 1 year), non-lactating, or of childbearing potential for whom a urine pregnancy test is negative when taken within the 24 h before administration of 89Zr-DFO-nimotuzumab.
* WHO performance status of 0 - 2
* Patients naïve to anti-EGFR antibodies treatment.

Exclusion Criteria:

* Unable to tolerate 60 min of PET imaging per session.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The observation of differences in 89Zr-DFO-nimotuzumab uptake between the tumors and normal tissues using PET/CT. | baseline (infusion) to day 7

SECONDARY OUTCOMES:
Lesion detection rate of FDG PET/CT compared with 89Zr-DFO-nimotuzumab in patients with EGFR-positive (by IHC) lung and colorectal cancers using PET/CT. | baseline (infusion) to day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No